CLINICAL TRIAL: NCT03790280
Title: High Frequency Oscillation in Pediatric Epilepsy Surgery
Acronym: HFO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HFO1001
Record Dates: First submitted 2018-12-21; First posted 2018-12-31 (Actual); Results first posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Pediatric Epilepsy; Epilepsy Surgery; High Frequency Oscillation

STUDY DESIGN:
Intervention Model Description: Randomization into standard arm and the treatment arm in a 1:1 ratio.
Who Masked: Participant, Care Provider
Masking Description: A double-blinded randomized control trial including children with refractory focal epilepsy who undergo surgery with intra- or extra-operative electrocorticography. Surgery is tailored by HFOs and standard ECoG interpretation (spikes on intra-operative ECoG or seizure onset on extra-operative ECoG) (arm 1), or tailored by standard ECoG alone (arm 2).
  Informed consent will be obtained 1 to 7 days to up to 3 months prior to the day of surgery. Prior to surgery, the subject will be randomized into the cohort arms in a 1:1 ratio.
  Blinding of the clinical neurophysiologists and neurosurgeons for treatment allocation is not feasible because of the character of the intervention. Therefore, this is a double-blinded trial as subjects will be blinded to the cohort arm to minimize bias of the follow-up results. The treating neurologist will also be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Standard of Care PLUS HFO (Experimental): Surgery is tailored by HFOs and standard ECoG interpretation (spikes on intra-operative ECoG or seizure onset on extra-operative ECoG) (arm 1).
  Interventions: Diagnostic Test: HFO analysis
- Standard of Care (No Intervention): Surgery is tailored by standard ECoG alone (arm 2).

INTERVENTIONS:
Diagnostic Test: HFO analysis — We hypothesize that the strategy of incorporating HFO data to a standard ECoG-guided resection in pediatric epilepsy surgery will result in improved postoperative seizure outcome than the traditional approach.
  Arms: Standard of Care PLUS HFO

SUMMARY:
High Frequency Oscillation (HFO) on ElectroCorticoGraphy (ECoG) has been identified as a new biomarker for epileptogenic tissue. The purpose of this study is to see if epilepsy surgery guided by the combination of HFO on ECoG and standard clinical practice can result in a greater likelihood of seizure freedom, versus standard clinical practice alone, without HFOs.

DETAILED DESCRIPTION:
Intra-operative electrocorticography (ECoG), based on interictal spike and spike patterns, is performed to optimize delineation of the epileptogenic tissue in the operating room during epilepsy surgery. Similarly, extra-operative electrocorticography is often recorded over days to weeks with intracranial grids and depth electrodes, when the epileptogenic zone is not clearly localized with non-invasive studies and/or with intra-operative ECoG. Surgical resection following extra-operative ECoG is then "tailored' by the seizure onset zone as the gold standard.

High frequency oscillations have been identified as a more precise biomarker for epileptogenic tissue. The aim of this double-blind randomized surgical trial is to determine if HFO- tailored surgery combining HFOs and current standard of care, compared to current standard of care alone, will lead to a better seizure outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age 0-21 years
* Refractory focal epilepsy
* Planned resective epilepsy neurosurgery
* Includes intraoperative or extraoperative electrocorticography with grids
* Planned resective epilepsy surgery approved by institutional surgery board

Exclusion Criteria:

* Subjects undergoing non-resective neurosurgery
* Does not include intraoperative or extraoperative electrocorticography with grids
* Planned resective surgery is a hemispherectomy/hemispherotomy

Ages: 0 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care PLUS HFO | Standard of Care
Started | 8 | 9
Completed | 7 | 9
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care PLUS HFO | Standard of Care | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 7 | 13
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Gender: Female | 5 | 5 | 10
  Gender: Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 7 | 6 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 4 | 7 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Seizure-free Rate
Description: The primary outcome measure is the number of patients seizure-free after surgery in the treatment arm of combined HFO and standard of care, compared to the number of patients seizure-free in the control arm of standard of care alone, at 1 year after surgery.
Time Frame: 1 year after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care PLUS HFO | Standard of Care
Number analyzed (Participants) | 8 | 9
Participants
  Seizure Free at 1 year post surgery | 4 | 5
  Seizure Relapse at 1 year post surgery | 4 | 4

2. Secondary Outcome: Post-operative Complication
Description: Number of participants experiencing surgical complications
Time Frame: 1 year after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care PLUS HFO | Standard of Care
Number analyzed (Participants) | 7 | 9
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected post-operatively for up to 1 year.
Groups:
- Standard of Care PLUS HFO: The primary outcome measure is the number of patients seizure-free after surgery in the treatment arm of combined HFO and standard of care, compared to the number of patients seizure-free in the control arm of standard of care alone, at 1 year after surgery.
Arm/Group | Standard of Care PLUS HFO | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 1/8 | 0/9
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care PLUS HFO (N=8) | Standard of Care (N=9)
Subdural Hematoma (Injury, poisoning and procedural complications) | 1 (1) | NA — Perioperative unwitnessed fall resulted in left subdural hematoma requiring evacuation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-10-26): https://cdn.clinicaltrials.gov/large-docs/80/NCT03790280/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-26): https://cdn.clinicaltrials.gov/large-docs/80/NCT03790280/SAP_001.pdf